CLINICAL TRIAL: NCT02310984
Title: PICTURE Breast XS: Patient Information Combined for Local Therapy oUtcome Assessment in bREast Cancer - Cross-sectional
Acronym: PICTURE XS
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: UCL 13/0354; 14/LO/0428 (Other: HRA NRES Committee)
Record Dates: First submitted 2014-09-03; First posted 2014-12-08 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2016-10

CONDITIONS: Early-Stage Breast Carcinoma
Keywords: Early breast cancer; Lumpectomy; Breast conserving surgery; Radiotherapy; Cosmesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This project which is fully funded by the European Union FP7 Program is designed to pull together all the information we obtain from scans and x-rays to design a personalised 3-D digital model of each patient, their anatomy and disease. We can then use this as follows: as (i) an aid to surgical planning to enable objective clinical decision making (ii) a decision support tool to communicate the available treatment options to the patient and facilitate shared decision making and provision of personalised care and (iii) to enable standardised objective evaluation of the aesthetic outcome of the treatment procedures. This study aims to demonstrate the ability of the Virtual Physiological Human concept to empower breast cancer patients and assess the impact on their care and quality of life.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer to affect women in Europe, having a lifetime risk of 1 in 9. It is an increasingly treatable disease, and 10-year survival now exceeds 80%. The primary treatment for breast cancer is surgery, which may be used in conjunction with adjuvant therapies, such as chemotherapy and radiotherapy. Given the high breast cancer survival rate, many women will live for many years with the potentially disfiguring aesthetic consequences of their surgical and therapeutic treatment. A good aesthetic outcome is an important endpoint for breast cancer treatment and is closely related to psychosocial recovery and quality of life.

When a woman faces a breast cancer diagnosis, and surgery is proposed, several options are available. The decision as to which type of surgery to offer patients is largely subjective and based almost exclusively on the judgment and experience of the clinician. The cosmetic outcome of surgery is a function of many factors including tumour size and location, the volume of the breast, its density, and the dose and distribution of radiotherapy. In breast-conserving surgery, there is evidence that approximately 30% of women receive a suboptimal or poor aesthetic outcome; however there is currently no standardised method of identifying these women.

The PICTURE project aims to address these issues by providing objective tools, tailored to the individual patient, to predict the aesthetic outcome of local treatment. Using a combination of 3D photography and routinely acquired radiological images (i.e. mammography, ultrasound and MRI, when available), together with information about the tumour (size, location, shape etc.) we will develop techniques to biomechanically model the anatomy of the breast and the effect of surgical removal of cancerous tissue. This digital patient representation and associated predictive tools will enable alternative surgical strategies to be explored and the consequences of the available options, with respect to the appearance of the breast, to be visualised. This will aid communication with the patient of the type of breast surgery recommended by the surgeon, and will empower patients to take an active role in a shared decision making process.

The study will develop tools to enable the patient's aesthetic appearance after treatment to be objectively evaluated. Current techniques use subjective methods, such as assessment by an expert panel, or computer analysis of 2-dimensional photography to estimate, for instance, breast asymmetry. By adopting recent developments in low cost 3D photography and depth sensing technology, we will develop a standardised, reproducible analysis tool which will base the aesthetic outcome evaluation on both the 3-dimensional shape of the reconstructed breast and its volume. This will establish standardised quality assurance and evaluation procedures, enabling institutions across Europe to be compared and factors that have a positive or negative impact on surgical outcome identified.

In summary, the demonstrator created by the PICTURE project will integrate models of surgical techniques and treatment schemes, clinical patient data, multi-modal imaging and individualised models of patient anatomy to build a personalised, digital representation of the patient. The aim is for this to be used as an aid to surgical planning, via simulation of the cosmetic effects of breast conserving surgery, as a decision support tool to communicate the available options to the patient and to enable standardised evaluation and a safe outcome of the procedure. The demonstrator aims to empower patients and will have a direct impact on their care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women who have undergone breast conserving surgery for early breast cancer more than one year ago.
* Written informed consent obtained.

Exclusion Criteria:

* Unable to provide written informed consent.
* Younger than 18 years.
* Benign breast disease.
* Women who have had a mastectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have undergone breast conserving surgery for early breast cancer more than one year ago.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the factors that determine aesthetic outcome after treatment for early breast cancer | Single assessment on one day, beyond one year from date of primary surgery.
  The primary aim of this study is to evaluate the factors that determine aesthetic outcome after treatment for early breast cancer, based on a consensual classification obtained with a consensus panel. The information thus obtained will be integrated into the demonstrator (a personalised digital representation of the patient).

SECONDARY OUTCOMES:
Comparison of the characteristics of this patient group with the group used to make the demonstrator in PICTURE L (composite outcome). | Single assessment on one day, beyond one year from date of primary surgery.
  Comparison of the characteristics of the primary tumour in this patient group with the group used to make the demonstrator. The characteristics include: primary tumour side, quadrant, size, and hormone receptor status.
Comparison of the characteristics of this patient group with the group used to make the demonstrator in PICTURE L (composite outcome). | Single assessment on one day, beyond one year from date of primary surgery.
  Comparison of the characteristics of treatment received in this patient group with the group used to make the demonstrator. The characteristics include: details of surgery, chemotherapy, radiotherapy and adjuvant hormonal therapy.
Comparison of the characteristics of this patient group with the group used to make the demonstrator in PICTURE L (composite outcome). | Single assessment on one day, beyond one year from date of primary surgery.
  Comparison of the characteristics assessed by questionnaire of this patient group with the group used to make the demonstrator. The characteristics include: measures assessed by the questionnaires (EQ-5D-5L, QLQ-C30 & BR23, and BREAST-Q).

CONTACTS AND LOCATIONS:
Overall Officials: Mo Keshtgar, MB BS, FRCS, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (3):
- Leiden University Medical Center (LUMC), Leiden, Netherlands
- Champalimaud Cancer Center, Lisbon, Portugal
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All requests for data sharing will adhere to the UCL Surgical & Interventional Trials Unit (SITU) data sharing agreement policy. UCL Medical School is supportive of data sharing and will endeavour to assist in requests for data sharing. These data will be held at UCL on secure servers and will not be released to any third parties until the final study report has been published. All requests for access to the data will be formally requested through the use of a SITU data request form which will state the purpose, analysis and publication plans together with the named collaborators. All requests are dealt with on a case by case basis. All requests will be logged and those successful will have a data transfer agreement which will specify appropriate acknowledgement of the Royal Free Hospital, the sponsor, and funders.

REFERENCES:
- See also: EU FP7 website — http://cordis.europa.eu/project/rcn/106628_en.html